CLINICAL TRIAL: NCT00834938
Title: Long Term Effects of Bariatric Surgery on Diabetes: Comparison Between Patients With or Without Diabetes Recovery.
Brief Title: Comparison Between Patients With or Without Diabetes Recovery After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fernanda Maria Possidonio Filgueira Hirsch, UNICAMP
Other Study IDs: LIMED0005
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes; Bariatric Surgery; Obesity
Keywords: diabetes mellitus, type 2; Insulin resistance; bariatric surgery; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin; adiponectin; Cytokines; gastric bypass; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with DM2 undergoing RYGB with remission of DM2
  Interventions: Other: No intervention
- 2: Patients with DM2 undergoing RYGB without remission of DM2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bariatric surgery can lead to improvement or even resolution of type 2 diabetes in about 80% of patients submitted to Roux-en-Y gastric bypass (RYGP). Otherwise, many patients experienced no resolution of their diabetes despite massive surgical-induced weight loss. There appears to be a variable response to surgery depending on surgical and patient factors. To explore potential factors affecting diabetes outcomes after RYGP, this study is proposed to make a description of effects of surgical procedures on incretin, insulin production and sensitivity and a comparison between patients with or without remission of Type 2 Diabetes.

DETAILED DESCRIPTION:
Diabetes reversion is observed after bariatric surgeries even before significant weight loss could explain it, mainly in predominantly malabsorptive procedures (98,9% for biliopancreatic diversion or duodenal switch), followed by those combining malabsorption and gastric restriction (83,7% for Roux-en-Y gastric bypass). Changes in the hormonal communication between the digestive system and the pancreas would explain the antidiabetogenic role of the surgery, so this effect could be obtained in nonobese, diabetic individuals.

To explore potential factors affecting diabetes outcomes after RYGP, this study is proposed to make a description of effects of surgical procedures on incretin, insulin production and sensitivity and a comparison between patients with or without remission of Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to understand the procedures of the study.
* To agree voluntarily to participate of the study, signing an informed consent.
* Weight variance less than 5% in the last 3 months.
* Operative group with at least 2 year follow-up.

Exclusion Criteria:

* History of hepatic disease like cirrhosis or chronic active hepatitis.
* Kidney dysfunction (creatinine > 1,4 mg/dl in women and > 1,5 mg/dl in men).
* Hepatic dysfunction: ALT and/or AST 3x above upper normal limit).
* Recent history of neoplasia (< 5 years).
* Use of oral or injectable for more than consecutive 14 days in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with DM2 and obesity undergoing RYGB with remission of DM2 and without remission.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Describe the endogenous response of incretins, orexins and anorexins to a mixed meal test in obese patients with DM2, in patients with DM2 undergoing RYGB with remission of DM2 and in patients without remission. | 2 years after RYGB

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Pareja, MD, PhD, Principal Investigator — University of Campinas, Brazil; Bruno Geloneze, MD, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Geloneze B, Tambascia MA, Pilla VF, Geloneze SR, Repetto EM, Pareja JC. Ghrelin: a gut-brain hormone: effect of gastric bypass surgery. Obes Surg. 2003 Feb;13(1):17-22. doi: 10.1381/096089203321136539. PMID 12630608
- [Background] Geloneze B, Tambascia MA, Pareja JC, Repetto EM, Magna LA. The insulin tolerance test in morbidly obese patients undergoing bariatric surgery. Obes Res. 2001 Dec;9(12):763-9. doi: 10.1038/oby.2001.105. PMID 11743060
- [Background] Pories WJ, MacDonald KG Jr, Flickinger EG, Dohm GL, Sinha MK, Barakat HA, May HJ, Khazanie P, Swanson MS, Morgan E, et al. Is type II diabetes mellitus (NIDDM) a surgical disease? Ann Surg. 1992 Jun;215(6):633-42; discussion 643. doi: 10.1097/00000658-199206000-00010. PMID 1632685
- [Background] Pories WJ. Diabetes: the evolution of a new paradigm. Ann Surg. 2004 Jan;239(1):12-3. doi: 10.1097/01.sla.0000102990.47956.98. PMID 14685094